CLINICAL TRIAL: NCT02792296
Title: A Study to Assess the Feasibility of and to Characterize Project: EVO Monitor Cognitive Function Measurements When Played Daily, Weekly, or Multiple Times Per Day in Adults 40-55 Years Old
Brief Title: Feasibility & Characterization of Project: EVO Monitor Cognitive Measurements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Akili-026
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daily measurement (Experimental): This arm will be asked to use the Project: EVO Monitor once a day for four weeks..
  Interventions: Other: Project: EVO Monitor
- Multiple times per day measurement (Experimental): This arm will be asked to use the Project: EVO Monitor at least once per day and six times over the day every three days for four weeks.
  Interventions: Other: Project: EVO Monitor
- Weekly measurement (Experimental): This arm will be asked to use the Project: EVO Monitor once a week for eight weeks.
  Interventions: Other: Project: EVO Monitor

INTERVENTIONS:
Other: Project: EVO Monitor — Project: EVO Monitor was designed to incorporate a proprietary multi-tasking assessment into a state-of-the-art mobile video game-like platform, which deploys modern videogame graphics, engaging reward loops, and real-time adaptive mechanics to dynamically personalize difficulty in order to assess the user's ability.

SUMMARY:
This is an open-label study in adults to assess at-home Project: EVO Monitor measurements over repeat play cycles. The study has three arms:playing multiple times per day, once daily, and once weekly for 4 to 8 weeks.

DETAILED DESCRIPTION:
This is an open-label study in adults ages 40 to 55 to assess Project: EVO Monitor measurements over repeat play cycles. The study has three arms: adults playing multiple times per day, adults playing once daily, and adults playing once weekly. The investigators plan to evaluate 76 participants (N = 30 in the daily and weekly arms, and N=16 in the multiple times per day arm) in two sites over a 4 to 8 week study period. The study period includes 2 in-clinic sessions and scheduled, at-home game play of the short (less than 7 minutes) Project: EVO Monitor.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-55 at the time of informed consent
* Ability to follow written and verbal instructions (English).
* Male and Female (Gender-matched).
* Ability to comply with all the testing and requirements.

Exclusion Criteria:

* Current, controlled (requiring a restricted medication) or uncontrolled, self-reported psychiatric diagnosis with significant symptoms such as post-traumatic stress disorder, psychosis, bipolar illness, pervasive developmental disorder, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder, conduct disorder, attention deficit disorder, autism spectrum disorder, or other symptomatic manifestations that in the opinion of the Investigator that may confound study data/assessments.
* Current self-reported community diagnosis of cognitive ailments such as dementia, Alzheimer's disease, stroke, traumatic brain injury, or other diseases that in the opinion of the Investigator that may confound study data/assessments.
* Current diagnosis of severe learning disorder, dyslexia, or dyscalculia.
* Current subjective complaints of inattention or memory loss.
* Current use of psychotropic medication, prescription or otherwise.
* Currently undergoing psychotherapy, behavioral therapy, or occupational therapy.
* Motor condition that prevents game playing, as observed by investigator.
* Impaired visual acuity, as defined by difficulty reading the informed consent even with corrective lenses.
* Recent history (within the past 6 months) of suspected substance abuse or dependence.
* History of seizures (exclusive of febrile seizures), a tic disorder, significant tics, a current diagnosis of Tourette's Disorder.
* Taken part in a clinical trial within 30 days prior to screening.
* Diagnosis of color blindness.
* Regular use of psychoactive drugs that in the opinion of the Investigator may confound study data/assessments
* Any other medical condition that in the opinion of the investigator may confound study data/assessments.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of at-home use as measured by percent of completed assigned sessions | 4 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ted Riley, Study Director — Promedica International
Locations (2):
- United States (2):
  - Preferred Research Partners, Little Rock, Arkansas
  - Clinical Trials of Texas, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No